CLINICAL TRIAL: NCT01644669
Title: A Safety and Efficacy Study of Intra-Operative Radiation Therapy (IORT) Using the Xoft® Axxent® eBx® System® at the Time of Breast Conservation Surgery for Early Stage Breast Cancer
Brief Title: Safety and Efficacy Study of the Xoft® Axxent® eBx® IORT System®
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Collaborators: Icad, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTPR-0009
Record Dates: First submitted 2012-06-28; First posted 2012-07-19 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Invasive Ductal Carcinoma; Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Intervention Model Description: Single 20Gy dose of electronic brachytherapy (IORT)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-operative Radiation Therapy - IORT (Experimental): Intra-operative Radiation Therapy
  Interventions: Radiation: Intra-operative Radiation Therapy - IORT

INTERVENTIONS:
Radiation: Intra-operative Radiation Therapy - IORT — Single dose of 20 Gy
  Other Names: Electronic Brachytherapy

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of the Xoft Axxent eBx System when used for single-fraction IORT in early stage breast cancer. Hypothesis: IORT using the Xoft Axxent eBx System is no worse (non-inferior) than whole breast irradiation (WBI) when used as stand-alone radiation treatment in breast conserving therapy in women with early stage breast cancer.

DETAILED DESCRIPTION:
The rationale for IORT as the sole radiation therapy is:

Favorable preliminary results in feasibility, safety and efficacy outcomes: Accelerated Partial Breast Irradiation (APBI) is an accepted alternative to whole breast irradiation following breast-conserving surgery for early stage breast cancer. Intra-Operative Radiation Therapy (IORT) is a form of APBI that allows radiation to be delivered directly to the open tumor bed following Breast Conservation Surgery (BCS). After 4 years of follow-up, IORT has shown equivalent disease control rates as whole breast irradiation.

Direct and timely radiation to the tumor bed: Radiation is delivered at to the target tissue (adjacent to the resection margins at the time of lumpectomy). It avoids treatment delays and eliminates weeks or months of post-surgical radiation therapy during which residual cancer cells might proliferate. An in vitro study showed that un-irradiated wound fluid stimulated the growth of breast cancer cells while irradiated wound fluid did not. Each month of delay in radiation treatment is associated with a 1% increase in the recurrence rate. Huang, et al., found a 5.8% recurrence rate in patients who received WBRT within 8 weeks of BCS compared with a 9.1% recurrence rate in patients who started radiotherapy 9-16 weeks after BCS.

Increased patient treatment compliance compared to conventional radiation therapy: Suitable early stage breast cancer patients are able to complete their breast cancer radiotherapy treatment at the time of BCS, which offers a convenient and potentially life-saving benefit to patients who might otherwise omit radiation therapy if it required lengthy travel or time commitments. In addition, healthcare resources, including both personnel and facilities, will be conserved by eliminating the overhead cost of multiple patient visits, eliminating waiting time for patients, and consolidating therapy to one visit combined with the surgical procedure.

Available Technology: The Xoft Axxent controller, x-ray source, and balloon applicator are cleared by the United States Food and Drug Administration (FDA) to deliver brachytherapy treatments using high dose rate x-ray radiation. The Xoft Axxent System has been used to treat breast cancer subjects using a multi-fraction APBI technique on an outpatient basis as part of two multi-center studies. The Xoft Axxent System enables the Radiation Oncologist to administer electronic brachytherapy without the use of a radioactive isotope in minimally shielded rooms. Characteristics of the Xoft System that make it well-suited for IORT include its portability and low energy photons, allowing for minimal shielding during the radiation therapy.

This protocol has been developed to further study the use of the Xoft Axxent eBx System in the delivery of IORT for subjects with early-stage breast cancer. The Xoft Axxent eBx System will be used according to the United States Food and Drug Administration (FDA) 510(k) cleared labeling; therefore, the use of the technology in this study is considered on-label and within the scope of the FDA cleared indication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have provided written Informed Consent
2. Subject must have biopsy-proven invasive ductal carcinoma or ductal carcinoma in situ of the breast
3. Subject must be female ≥ 40 years of age
4. Subject's tumor(s) must be < 3.0 cm in greatest diameter by pre-operative assessment
5. Subject's tumor(s) must meet AJCC Tumor Classification: Tis, T1 or T2 (< 3 cm), N0, M0
6. Subject presenting with bilateral breast cancer may be enrolled if BOTH cancers meet all of the inclusion and none of the exclusion criteria
7. Women of child-bearing potential must have a negative pregnancy test within one week of IORT treatment
8. Women of child-bearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives or a combination of condom and spermicide) from the time of negative pregnancy test through completion of the radiation treatment period

Exclusion Criteria:

1. Subject is pregnant or nursing
2. Subject has significant auto-immune disease
3. Subject has a pacemaker present in the field of radiation or quadrant of the breast cancer
4. Subject has biopsy-proven multifocal breast cancer
5. Subject has multi-centric breast cancer
6. Subject has known lympho-vascular invasion
7. Subject has invasive lobular cancer
8. Subject has undergone neo-adjuvant chemotherapy or neo-adjuvant endocrine therapy for current breast cancer
9. Subject has a history of recurrent breast cancer in the ipsilateral breast
10. Subject has had previous radiation exposure of the involved breast
11. Subject has BRCA 1 or 2 mutations. Note: Testing will only be required for Subjects presenting with bilateral breast cancer; testing is not required for unilateral cancers
12. Subject has contraindications for radiation
13. Subject considered by the Investigator to be high-risk for breast conservation surgery and/or intra-operative radiation therapy
14. Subject has participated in any other clinical investigation that is likely to confound study results or affect study outcome either at the time of IORT or for 3 months prior to IORT.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-05-08 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the rate of ipsilateral breast tumor recurrence (IBTR) at 5 years | Change from baseline reported at 5 years
  IBTR is defined as biopsy-proven reappearance of cancer in the treated breast. IBTR will be assessed at Month 6, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. A non-inferiority comparison to whole breast irradiation will be made at 5 years.

SECONDARY OUTCOMES:
Assess the rate of regional breast tumor recurrence (RBTR) | Report at 10 yrs
  Regional breast tumor recurrence is defined as biopsy-proven reappearance of cancer in the axilla. Regional recurrence will be assessed at Month 6, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. Regional recurrence rates will be compared to the historical control of WBI at 5 and 10 years.
Disease Free Survival Rate (DFSR) and Overall Survival rate | Report at 5 and 10 years
  Disease free survival (DFS) is defined as the length of time from IORT to any first recurrence. The incidence of disease free survival will be assessed at Month 1, Month 6, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. DFS will be compared to the historical control at 5 and 10 years.
Cosmetic Outcome | Report at 5 and 10 yrs
  Cosmetic outcome will be recorded at baseline, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. a. Physician evaluation will be done using the Harvard Scale.
Quality of Life (QOL) | Reported at 5 and 10 yrs
  Quality of Life will be assessed at baseline and at each follow-up visit: Month 1, Month 6, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. QOL will be measured using the FACT-B self-reporting questionnaires.
Assess the safety of single fraction IORT at the time of breast conserving surgery for early stage breast cancer | On-going monitoring, report at 5 and 10 years
  The rates and severity of Adverse Events (AEs), Adverse Device Effects (ADEs), and Unanticipated Adverse Device Effects (UADEs) during and following IORT will be assessed at each follow-up visit. Safety events will be compared to the historical control of WBI at 5 and 10 years. Each event will be classified according to the following: Device Related, Procedure Related or Radiation Related.
Assess the rate of ipsilateral breast tumor recurrence (IBTR) at 10 years | Change from baseline reported at 10 years
  IBTR is defined as biopsy-proven reappearance of cancer in the treated breast. IBTR will be assessed at Month 6, Month 12, Month 18, Year 2, and then annually through ten (10) year follow-up. A non-inferiority comparison to whole breast irradiation will be made at 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: A.M. Nisar Syed, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (24):
- United States (22):
  - University of Arizona, Tucson, Arizona
  - City of Hope, Duarte, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - UCLA, Los Angeles, California
  - Tri-City Medical Center, Oceanside, California
  - Diablo Valley Oncology Hematology Medical Group, Pleasant Hill, California
  - Western Surgical Care, PC, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Florida Hospital Celebration Health, Celebration, Florida
  - Doctors Hospital, Coral Gables, Florida
  - Martin Health System Center for Clinical Research, Stuart, Florida
  - Rush University, Chicago, Illinois
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Oncology Network - Good Samaritan Hospital, Baltimore, Maryland
  - MedStar Oncology Network - Franklin Square, Baltimore, Maryland
  - Exeter Hospital, Exeter, New Hampshire
  - Staten Island University Hospital, Staten Island, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Sentara Northern Virginia Medical Center, Woodbridge, Virginia
- Monash Health / Peter MacCallum Cancer Centre, Clayton, Victoria, Australia
- Hospital CUF Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Ivanov O, Dickler A, Lum BY, Pellicane JV, Francescatti DS. Twelve-month follow-up results of a trial utilizing Axxent electronic brachytherapy to deliver intraoperative radiation therapy for early-stage breast cancer. Ann Surg Oncol. 2011 Feb;18(2):453-8. doi: 10.1245/s10434-010-1283-x. Epub 2010 Aug 25. PMID 20737219
- [Background] Dickler A, Ivanov O, Francescatti D. Intraoperative radiation therapy in the treatment of early-stage breast cancer utilizing xoft axxent electronic brachytherapy. World J Surg Oncol. 2009 Mar 2;7:24. doi: 10.1186/1477-7819-7-24. PMID 19254369
- See also: National Cancer Institute Factsheet - Radiation Therapy for Cancer — http://www.cancer.gov/cancertopics/factsheet/Therapy/radiation